CLINICAL TRIAL: NCT01496378
Title: Problem Solving Skills Training For Parent Caregivers of Youth With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HD065180-01A1 (NIH)
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Chronic Pain; Abdominal Pain; Headache
Keywords: Chronic Pain; Abdominal Pain; Headache; Adolescents; Children; Parents; Problem-Solving Skills Training
MeSH Terms: conditions — Chronic Pain; Abdominal Pain; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem-Solving Skills Training (Experimental): In addition to standard medical care, parents in the problem-solving skills training group will receive 8 sessions (1 hour each) of individual problem-solving therapy over 8 weeks. Caregivers will be asked to complete the first training session and at least 3 subsequent sessions in person at their local treatment facility (Seattle Children's Hospital or Oregon Health and Science University). Remaining sessions will be completed via telephone.
  Interventions: Behavioral: Problem-Solving Skills Training
- Standard Care (No Intervention): Parents and children in the Standard Care group will continue with the care that has been prescribed for their child's pain problem by their treating physician, which may include medications, physical therapy, and mental health intervention.

INTERVENTIONS:
Behavioral: Problem-Solving Skills Training — Parents will receive 8, 1-hour sessions of individual problem-solving therapy over 8 weeks. Caregivers will complete the first training session and at least 3 subsequent sessions in person. Remaining sessions will be completed via telephone. In session 1, parents will be introduced to the PSST program and a rationale and explanation for problem solving strategies will be provided. During sessions 2-8, parents will identify a problem that they wish to work on. The therapist will use the primary cognitive-behavioral strategies of modeling, behavioral rehearsal, performance feedback, and generalization of skills in the process of teaching problem solving skills to parents. Parents will complete homework assignments to practice using the problem-solving skills in real-life situations
  Arms: Problem-Solving Skills Training

SUMMARY:
The purpose of this study is to evaluate the feasibility and efficacy of problem-solving skills training (PSST) to reduce distress and increase coping abilities among parents of youth with chronic pain. We hypothesize that parents will complete the PSST intervention and will find it to be an acceptable and satisfactory treatment. We also hypothesize that parents who receive PSST will have less distress and better coping skills than parents who receive standard care, and that children of parents who receive PSST will have better physical and emotional functioning than children of parents who receive standard care.

DETAILED DESCRIPTION:
Chronic pain affects 25-40% of children and adolescents, and results in significantly lower quality of life for these youth. Parents play an important role in how their children cope with chronic pain, and can also experience their own distress related to their child's illness. Parental psychological distress is widely recognized to be associated with poorer child adjustment. However, no interventions have been developed specifically to treat psychological distress in parents of children with chronic pain. Problem-solving skills training (PSST) has been shown to result in significant reductions in parental distress among caregivers of children with other types of chronic illness such as cancer. The purpose of this study is to test the feasibility and preliminary efficacy of PSST for parents of youth with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Child age 10-17 years
* Child's pain present for at least 3 months duration
* Pain occurs at least 1 time per week and interferes with daily functioning
* Pain is not related to a chronic disease
* Receiving evaluation or treatment in a pediatric pain clinic
* Literate in English

Exclusion Criteria:

* A serious comorbid chronic condition in the child (e.g., diabetes, arthritis, cancer)
* Non-English speaking
* Parent has lived with the child for less than one year
* Parent has active psychosis or suicidal ideation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in problem solving skills from baseline to immediately post-treatment and 3-month follow-up | baseline, immediately post-treatment, 3-month follow-up
  Parent report of problem solving skills will be assessed using the Social Problem Solving Skills Inventory-Revised, which includes 52 items consisting of 5 scales that measure 2 different problem orientation dimensions (Positive and Negative) and three different problem-solving proper dimensions (Irrational Problem-Solving, Impulsivity/Carelessness Style, and Avoidance style).
Change in depressive symptoms from baseline to immediately post-treatment and 3-month follow-up | baseline, immediately post-treatment, 3-month follow-up
  Parents will complete the Beck Depression Inventory-II (BDI-II) to assess parental depressive symptoms. The BDI-II is a 21-item measure that assesses the cognitive, affective, and behavioral components of depressive symptoms in adults.
Change in anxiety and depressive symptoms from baseline to immediately post-treatment and 3-month follow-up | baseline, immediately post-treatment, 3-month follow-up
  Parents will complete the Profile of Mood States (POMS) to assess parent anxiety and depressive symptoms. The POMS is a 30-item measure that asks about feelings over the previous week. Six affective states are assessed: tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. These subscales are combined to form a total POMS score.
Change in parenting stress from baseline to immediately post-treatment and 3-month follow-up | baseline, post-treatment, 3-month follow-up
  Parents will complete the Parenting Stress Index-Short Form(PSI-SF) to assess parenting stress. The PSI-SF is a 36-item questionnaire that assesses parental distress, parent-child dysfunctional interactions, and difficulty parenting.
Change in child physical and emotional functioning from baseline to immediately post-treatment and 3-month follow-up | baseline, post-treatment, 3-month follow-up
  Children will complete the Bath Adolescent Pain Questionnaire (BAPQ), a 61-item measure that measures the impact of pain on child physical and emotional functioning. The BAPQ was developed specifically for children with chronic pain. Subscales measuring children's depression and physical functioning will be used in analyses.

SECONDARY OUTCOMES:
Change in parental impact of chronic pain from baseline to immediately post-treatment and 3-month follow-up | baseline, immediately post-treatment, and 3-month follow-up
  Parents will complete the Bath Adolescent Pain Questionnaire-Parent Impact to assess changes in functioning and behavior associated with parenting an adolescent with chronic pain. This is a 62-item scale. Two subscales will be used in analyses: child-related catastrophizing and parental behavior.
Treatment expectancies | baseline
  Parents will complete a 10-item treatment expectancies questionnaire to rate the likelihood that treatment will lead to symptom improvement on a 5-point rating scale (0="not at all likely" to 4="extremely likely").
Brief symptom inventory | baseline
  Parents will complete the Brief Symptom Inventory, an 18-item questionnaire that assesses parental general psychological distress.
Treatment satisfaction | immediately post-treatment and 3-month follow-up
  Parents will complete an 8-item scale regarding satisfaction with the therapeutic process during the course of treatment and satisfaction with the outcome of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya M. Palermo, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - Seattle Children's Hospital, Seattle, Washington